CLINICAL TRIAL: NCT01420276
Title: Female Sexual Function and Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Bezmialem Vakif University, Bezmialem Vakif University
Other Study IDs: gbpk1
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Female Sexual Function
Keywords: Female sexual function

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Back paın is a common hormonal disorder in women that may affect the phases of female sexual function (FSD). We investigated sexual function in patients with back paın A total of 54 women with back paın and 27 age matched voluntary healthy women who served as the as control group were evaluated with a detailed medical and sexual history, including a female sexual function index (FSFI) questionnaire and the Beck Depression Inventory. Serum prolactin, dehydroepiandrosterone sulfate, free testosterone, androstenedione, 17alpha-hydroxyprogesterone, estradiol, free thyroxin and thyrotropin were measured. These variables were compared statistically between the 2 groups.

DETAILED DESCRIPTION:
A total of 54 women with back paın and 27 age matched voluntary healthy women who served as the as control group were evaluated with a detailed medical and sexual history, including a female sexual function index (FSFI) questionnaire and the Beck Depression Inventory. Serum prolactin, dehydroepiandrosterone sulfate, free testosterone, androstenedione, 17alpha-hydroxyprogesterone, estradiol, free thyroxin and thyrotropin were measured. These variables were compared statistically between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 year old
* Female
* Active sexual life

Exclusion Criteria:

* Younger than 20, older than 45 year old.
* Menopause

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female with active sexual life
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Female sexual function | 6 months